CLINICAL TRIAL: NCT04070430
Title: Crutch Use After Arthroscopic Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-01106
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Hip Fractures; Hip Injuries
Keywords: Arthroscopic hip surgery
MeSH Terms: conditions — Hip Fractures; Hip Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 weeks of partial weight bearing on crutches (Active Comparator): post-operative patient reported outcome (PRO) scores will be collected 6 weeks, 6 months, 12 months, and 24 months post-operatively
  Interventions: Other: 2 weeks of partial weight bearing on crutches
- 4 weeks of partial weight bearing on crutches (Active Comparator): post-operative patient reported outcome (PRO) scores will be collected 6 weeks, 6 months, 12 months, and 24 months post-operatively
  Interventions: Other: 4 weeks of partial weight bearing on crutches

INTERVENTIONS:
Other: 2 weeks of partial weight bearing on crutches — Following surgery, patients will be instructed by their surgeon to use crutches for 2 weeks, and will follow-up normally, as any patient would. Their crutch use will not impact the quality or style of their postoperative care in any manner. At their 6-week, 6-month, 12-month, and 24 months postoperative visit, the mHHS and NAHS scores will be collected and stored in a secure data system, REDCAPS.
  Arms: 2 weeks of partial weight bearing on crutches
Other: 4 weeks of partial weight bearing on crutches — Following surgery, patients will be instructed by their surgeon to use crutches for 4 weeks, and will follow-up normally, as any patient would. Their crutch use will not impact the quality or style of their postoperative care in any manner. At their 6-week, 6-month, 12-month, and 24 months postoperative visit, the mHHS and NAHS scores will be collected and stored in a secure data system, REDCAPS.
  Arms: 4 weeks of partial weight bearing on crutches

SUMMARY:
The purpose of this study is to determine whether crutch use for 4 weeks following hip arthroscopic surgery is superior to crutch use for 2 weeks following hip arthroscopic surgery. The primary objective of the study is to compare PRO scores between patients who have used crutches for 2 weeks and patients who have used crutches for 4 weeks.

DETAILED DESCRIPTION:
This will be a single-center, randomized prospective study. The study will compare post-operative patient reported outcome (PRO) scores including the modified Harris hip score (mHHS) and the non arthritic hip score (NAHS), both are externally-validated surveys for hip function. One cohort will be assigned a rehabilitation regimen that includes 2 weeks of partial weight bearing on crutches, and the other will be assigned a regimen of 4 weeks of partial weight.

ELIGIBILITY:
Inclusion Criteria:

* Hip arthroscopic surgery

Exclusion Criteria:

* Any surgery other than hip arthroscopy
* Age: less than 18 years of age
* Age: greater than 64 years of age
* Pregnant patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Change in patient-reported-outcome (PRO) survey | 6 weeks, 6 months, 12 months, and 24 months post-operatively.
Change in modified Harris hip score (mHHS) | 6 weeks, 6 months, 12 months, and 24 months post-operatively.
Change in Non arthritic hip score (NAHS) | 6 weeks, 6 months, 12 months, and 24 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Youm, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.

REFERENCES:
- [Derived] Shankar DS, Mojica ES, Blaeser AM, Vasavada KD, Bi AS, Youm T. Crutch use for 4 weeks vs. 1 week after hip arthroscopy for femoroacetabular impingement: A pseudorandomized clinical trial with 6-month follow-up. Bull Hosp Jt Dis (2013). 2025 Dec 1;83(1):129-134. doi: 10.1097/bh9.0000000000000020. Epub 2025 Dec 3. PMID 41637607